CLINICAL TRIAL: NCT07125079
Title: Blood-based Biomarkers of Acute Lung Injury/Acute Respiratory Distress Syndrome
Brief Title: Lung Injury is One of the Primary Causes of Morbidity and Mortality in Critically Ill Patients. These Patients Will be Monitored for: 1) Immune Cell Activation 2) Blood-based Biomarkers. In Vitro Models Derived From These Samples Will be Treated With Novel Agent PIP-2 to Evaluate Its Efficacy.
Acronym: ALI/ARDS
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Peroxitech Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: Biomarkers of Lung Injury
Record Dates: First submitted 2025-05-30; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: ROS; ARDS; PIP-2; immune cells; peripheral blood mononuclear cells
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with ARDS

SUMMARY:
Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS) is a condition where high levels of inflammation damage the lung. This is a highly morbid condition with no specific pharmacologic therapies. The investigators posit that ARDS is caused due to an exaggerated activation of immune cells and that blockade of this activation may reduce lung damage/injury and help in ARDS management and possibly recovery. To test this hypothesis, the investigators propose to generate an in vitro immune cell model and test a novel (reactive oxygen species) blocking agent PIP-2 on this model. The investigating team will obtain blood of ARDS patients and isolate immune cells (specifically peripheral blood mononuclear cells or PBMC) and monitor the activation of these cells and their blockade by PIP-2. This is entirely an in vitro study.

DETAILED DESCRIPTION:
The research study is being conducted to understand the behavior of immune cells in a patient with Acute Respiratory Distress Syndrome (ARDS). Immune cells protect humans from external threats like infection. However, if these cells are overactive, they can lead to an infection progressing into ARDS. ARDS arises as a result of extensive damage possibly due to overactivated immune cells. This project aims to understand the link between immune cell activation and ARDS.

To do so, the investigators will isolate immune cells specifically peripheral blood mononuclear cells (PBMC) from blood of ARDS patients. These cells will be utilized for in vitro experiments by checking for overactivation. Cells in vitro will also be treated with a novel synthetic agent PIP-2 (being developed Peroxitech Inc. a Collaborator of this study) to check if PIP-2 can reduce overactivation as monitored by the production of reactive oxygen species.

ELIGIBILITY:
Inclusion Criteria: ARDS patients with mild and moderate to severe ARDS. This will be based on PaO2/FiO2 in the range of 100 mmHg (severe) and moderate (100-200 mm Hg) and mild (200-300 mm Hg) -

Exclusion Criteria: Pregnant women, children will be excluded.

-

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Hospital Of the University of Pennsylvania at the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Reactive oxygen species in vitro | From enrollment until 21 days
  Peripheral Blood Mononuclear cells (PBMC) isolated

CONTACTS AND LOCATIONS:
Overall Officials: Shampa Chatterjee, PhD, Principal Investigator — University of Pennsylvania; Christian Bermudez, MD, Principal Investigator — University of Pennsylvania; Asad Usman, MD, Study Director — University of Pennsylvania
Locations (1):
- Hospital Of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT07125079/Prot_SAP_000.pdf